CLINICAL TRIAL: NCT05453903
Title: A Phase 1b Study of Bleximenib in Combination With AML-Directed Therapies for Participants With Acute Myeloid Leukemia Harboring KMT2A or NPM1 Alterations
Brief Title: A Study of Bleximenib in Combination With Acute Myeloid Leukemia (AML) Directed Therapies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109124; 75276617ALE1002 (Other: Janssen Research & Development, LLC); 2021-003999-14 (EudraCT Number); 2023-506582-58-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-07-08; First posted 2022-07-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine; Cytarabine; Daunorubicin; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Relapsed/Refractory Setting (Experimental): Participants with relapsed/refractory AML harboring NPM1, KMT2A, NUP98, or NUP214 alterations will receive bleximenib in combination with either venetoclax (VEN) (Cohort A1: bleximenib+VEN) or azacitidine (AZA) (Cohort A2: bleximenib +AZA) or VEN+AZA (Cohort A3: bleximenib+VEN+AZA) or VEN + AZA (Cohort A4: bleximenib + VEN + AZA) in adolescent participants aged greater than or equal to (>=) 12 years and less than (<) 18 years of age, to select the recommended phase 2 dose (RP2D) of bleximenib in combination with VEN, AZA or VEN+AZA (dose selection). In dose expansion portion of the study, participants will receive bleximenib in combination with AML directed therapies at the RP2D(s).
  Interventions: Drug: Bleximenib; Drug: Venetoclax (VEN); Drug: Azacitidine (AZA)
- Arm B: Newly Diagnosed Chemotherapy Ineligible Setting (Experimental): Participants will receive bleximenib in combination with VEN+AZA as frontline chemo therapy for newly diagnosed AML participants harboring KMT2A, NPM1, NUP98, or NUP214 alterations who are >=75 years of age or >=18 years of age to <75 years of age with comorbidities that preclude the use of intensive induction chemotherapy.
  Interventions: Drug: Bleximenib; Drug: Venetoclax (VEN); Drug: Azacitidine (AZA)
- Arm C: Newly Diagnosed Chemotherapy Eligible Setting (Experimental): Participants will receive combination of bleximenib with cytarabine+daunorubicin or idarubicin chemotherapy as frontline treatment regimen for participants >= 18 to <75 years of age with AML harboring NPM1, KMT2A, NUP98, or NUP214 alterations and eligible for intensive chemotherapy.
  Interventions: Drug: Bleximenib; Drug: Cytarabine; Drug: Daunorubicin or Idarubicin

INTERVENTIONS:
Drug: Bleximenib — Participants will receive bleximenib.
  Other Names: JNJ-75276617
Drug: Venetoclax (VEN) — Participants will receive VEN.
  Arms: Arm A: Relapsed/Refractory Setting; Arm B: Newly Diagnosed Chemotherapy Ineligible Setting
Drug: Azacitidine (AZA) — Participants will receive AZA.
  Arms: Arm A: Relapsed/Refractory Setting; Arm B: Newly Diagnosed Chemotherapy Ineligible Setting
Drug: Cytarabine — Participants will receive cytarabine.
  Arms: Arm C: Newly Diagnosed Chemotherapy Eligible Setting
Drug: Daunorubicin or Idarubicin — Participants will receive daunorubicin or idarubicin.
  Arms: Arm C: Newly Diagnosed Chemotherapy Eligible Setting

SUMMARY:
The purpose of this study is to determine the recommended Phase 2 dose (RP2D) candidate(s) of bleximenib in combination with AML directed therapies (dose selection) and further to evaluate safety and tolerability of bleximenib in combination with AML directed therapies at the RP2D(s) (dose expansion).

ELIGIBILITY:
Inclusion Criteria:

* Adolescent participants (defined as greater than or equal to [>=] 12 and less than [<] 18 years of age) are only eligible for the relapsed/refractory (R/R) cohort (Arm A, cohort A4)
* Diagnosis of AML according to World Health Organization (WHO) criteria: a) De novo or secondary AML; b) relapsed/refractory (Arm A only); c) harboring KMT2A, NPM1, NUP98, or NUP214 alterations; d) Participants may receive emergency leukapheresis and/or cytarabine as cytoreductive therapy according to local practice guidelines
* Pretreatment clinical laboratory values meeting the following criteria -listed below: White blood cell (WBC) count: less than or equal to (<=) 25*10^9 per liter (/L), adequate liver and renal function
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0, 1 or 2. Adolescent participants only: Performance status >70 by Lansky scale (for participants <16 years of age) or >70 Karnofsky scale (for participants >16 years of age)
* A female of childbearing potential must have a negative highly sensitive serum beta-human chorionic gonadotropin at screening and within 48 hours prior to the first dose of study treatment
* Must sign an informed consent form (ICF) indicating participant (or their legally authorized representative) understands the purpose of the study and procedures required for the study and is willing to participate in the study
* Willing and able to adhere to the prohibitions and restrictions specified in this protocol

Exclusion Criteria:

* Acute promyelocytic leukemia, diagnosis of Down syndrome associated leukemia or juvenile myelomonocytic leukemia according to WHO 2016 criteria
* Leukemic involvement of the central nervous system
* Recipient of solid organ transplant
* Cardiovascular disease that is uncontrolled, increases risk for Torsades de Pointes or that was diagnosed within 6 months prior to the first dose of study treatment including, but not limited to: (a) Myocardial infarction; (b) Severe or unstable angina; (c) Clinically significant cardiac arrhythmias, including bradycardia (<50 beats per minute); (d) Uncontrolled (persistent) hypertension: (example, blood pressure greater than [>] 140/90 millimeters of mercury [mm Hg]; (e) Acute neurologic events such as stroke or transient ischemic attack, intracranial or subarachnoid hemorrhage, intracranial trauma; (f) Venous thromboembolic events (example, pulmonary embolism) within 1 month prior to the first dose of study treatment ;(g) Congestive heart failure (NYHA class III to IV); (h) Pericarditis or clinically significant pericardial effusion; (i) Myocarditis; (j) Endocarditis (k) Clinically significant hypokalemia, hypomagnesemia, hypocalcemia (corrected for hypoalbuminemia)
* Any toxicity (except for alopecia, stable peripheral neuropathy, thrombocytopenia, neutropenia, anemia) from previous anticancer therapy that has not resolved to baseline or to grade 1 or less
* Pulmonary compromise that requires the need for supplemental oxygen use to maintain adequate oxygenation
* Participants with diagnosis of Fanconi anemia, Kostmann syndrome, Shwachman diamond syndrome, or any other known bone marrow failure syndrome

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-03-19 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 3 Years 3 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with Adverse Events (AEs) by Severity | Up to 3 Years 3 months
  Number of Participants with AEs by severity will be reported. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Number of Participants with Dose-limiting Toxicity (DLT) | End of Cycle 1 (28 days)
  Number of participants with DLT will be reported according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.

SECONDARY OUTCOMES:
Plasma Concentration of Bleximenib | Up to 3 Years 3 months
  Plasma samples will be analyzed to determine concentrations of bleximenib using a validated, specific, and sensitive method.
Number of Participants with Depletion of Leukemic Blasts | Up to 3 Years 3 months
  Number of participants with depletion of leukemic blasts will be reported.
Percentage of Participants who Achieve Complete Remission (CR) | Up to 3 Years 3 months
  Percentage of participants who achieve complete Remission (CR) will be reported. CR is defined as Bone marrow blasts less than (<) 5 percent (%); Absence of circulating blasts; Absence of extramedullary disease; Absolute neutrophil count (ANC) greater than or equal to (>=) 1.0*10^9/Liter (L) (1,000/microliter [mcL]); Platelet count >= 100 * 10^9/L (100,000/mcL).
Percentage of Participants who Achieve Complete Remission with Partial Hematologic Recovery (CRh) | Up to 3 Years 3 months
  Percentage of participants who achieve complete remission with partial hematologic recovery (CRh) will be reported. CRh is defined as All criteria of CR with both ANC >0.5 * 10^9/L (500/mcL) and platelet count >50 * 10^9/L (50,000/mcL).
Percentage of Participants who Achieve Complete Remission with Incomplete Hematologic Recovery (CRi) | Up to 3 Years 3 months
  Percentage of participants who achieve complete remission with incomplete hematologic recovery (CRi) will be reported. CRi is defined as All CR criteria except for residual neutropenia (<1.0*10^9/L [1,000/mcL]) or thrombocytopenia (<100 * 10^9/L [100,000/mcL]).
Percentage of Participants who Achieved Overall Response | Up to 3 Years 3 months
  Percentage of participants who achieve overall response will be reported. Overall response rate (ORR) is defined as the percentage of participants achieving CR, CRh, or CRi, morphologic leukemia-free state (MLFS) or partial remission (PR).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (32):
- United States (7):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Albert Einstein College Of Medicine, New York, New York
  - Novant Health, Charlotte, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - MD Anderson, Houston, Texas
- Australia (3):
  - Monash Medical Centre, Clayton
  - Peter MacCallum Cancer Centre, Melbourne
  - Westmead Hospital, Westmead
- Princess Margaret Cancer Centre University Health Network, Toronto, Ontario, Canada
- France (4):
  - Institut Paoli Calmettes, Marseille
  - Chu Rennes Hopital Pontchaillou, Rennes
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - CHU de Tours - Hôpital de Bretonneau, Tours
- Germany (5):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitatsklinikum Ulm, Ulm
- Italy (4):
  - Azienda Opedaliero-Universitaria Policlinico Sant'orsola Malpighi di Bologna, Bologna
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - IRCCS Istituto Clinico Humanitas, Rozzano
- Spain (5):
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Clinica Univ. de Navarra, Pamplona
- United Kingdom (3):
  - University College London Hospitals NHSFT, London
  - Christie Hospital NHS Trust, Manchester
  - Oxford University Hospitals NHS Trust, Oxfordshire

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Kwon MC, Thuring JW, Querolle O, Dai X, Verhulst T, Pande V, Marien A, Goffin D, Wenge DV, Yue H, Cutler JA, Jin C, Perner F, Hogeling SM, Shaffer PL, Jacobs F, Vinken P, Cai W, Keersmaekers V, Eyassu F, Bhogal B, Verstraeten K, El Ashkar S, Perry JA, Jayaguru P, Barreyro L, Kuchnio A, Darville N, Krosky D, Urbanietz G, Verbist B, Edwards JP, Cowley GS, Kirkpatrick R, Steele R, Ferrante L, Guttke C, Daskalakis N, Pietsch EC, Wilson DM, Attar R, Elsayed Y, Fischer ES, Schuringa JJ, Armstrong SA, Packman K, Philippar U. Preclinical efficacy of the potent, selective menin-KMT2A inhibitor JNJ-75276617 (bleximenib) in KMT2A- and NPM1-altered leukemias. Blood. 2024 Sep 12;144(11):1206-1220. doi: 10.1182/blood.2023022480. PMID 38905635